CLINICAL TRIAL: NCT06569186
Title: Cue-Based Vs. Clinician-Driven Feeding in Very Low Birthweight Infants: A Pilot Randomized Trial
Brief Title: Cue-Based Vs. Clinician-Driven Feeding in Very Low Birthweight Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012540
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Infant, Very Low Birth Weight; Infant Development; Feeding Patterns
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Intervention and Control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Cue-based feedings
  Interventions: Behavioral: Cue-based feedings
- Control (No Intervention): Clinician based feedings

INTERVENTIONS:
Behavioral: Cue-based feedings — Speech therapists will use cue-based protocols to guide feeds
  Other Names: Speech therapy driven feeds
  Arms: Intervention

SUMMARY:
In this parallel-group randomized controlled trial, very low birthweight infants will be randomly assigned in a 1:1 ratio to either cue-based (intervention group) or clinician-driven feeding (control group). For infants in the intervention group, Speech therapists and nurses will use their cue-based assessment training to aid in clinical management of oral feeding. For infants in the control group, clinicians caring for these infants will define the feeding plan based on their daily assessment.

ELIGIBILITY:
Inclusion criteria:

* Birthweight < 1500 grams
* Gestational age between 28 and 31 weeks of gestation
* Full enteral feeding established before 32 weeks of postmenstrual age (PMA)
* Oral feeding initiated before 33 weeks PMA.

Exclusion criteria:

* Major congenital/chromosomal anomalies,
* Patent ductus arteriosus causing significant cardiovascular symptoms
* History of necrotizing enterocolitis stage 2 or greater

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Time interval in days from introduction to attainment of independent oral feeding | 4-20 days

SECONDARY OUTCOMES:
Postnatal age at discharge in days | 34 to 40 weeks postnatal age
Length of hospital stay in days | 10-60 days
Average weight gain during the transition from tube to oral feeding | 10-60 days
Total number of tube feeding events per infant during the transition from tube to oral feeding | 10-60 days
Follow up phone call | 4-6 months after birth
  A follow-up phone call 3 months after NICU discharge will also be performed to assess long-term outcomes including the need for tube feeding or hospitalizations related to feeding/nutrition problems.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States